CLINICAL TRIAL: NCT03286244
Title: Safety and Preliminary Efficacy of CM082 in Combination With Paclitaxel for Treating Advanced Gastric Cancer Who Progressed on Standard First-line Treatment: a Phase 1, Dose-escalation Study
Brief Title: Second-line CM082 Combined With Paclitaxel For Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-104
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — vorolanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 plus paclitaxel (Experimental): In dose-escalation part, patients will be treated in dose levels at the following daily doses of CM082 and paclitaxel to establish the MTD and RP2D:
  CM082 100mg qd + paclitaxel 80mg/m2/day; CM082 150mg qd + paclitaxel 80mg/m2/day; CM082 200mg qd + paclitaxel 80mg/m2/day; In dose-expansion part, patients will be treated at the RP2D established in dose escalation part.
  Interventions: Drug: CM082 plus paclitaxel

INTERVENTIONS:
Drug: CM082 plus paclitaxel — CM082 treatment: A treatment cycle is defined as 28 days. Oral CM082 tablets was given once daily for 3 weeks followed by 1-week break with escalating dose (100 mg, 150 mg and 200mg).
  Drug: Paclitaxel Paclitaxel 80 mg/m2 will be administrated by intravenous injection on days 1, 8, 15 of a 28-day cycle for no more than 6 cycles.

SUMMARY:
This is an open-label, Phase 1b study which will be conducted in two parts: part A is the dose escalation study while part B is dose expansion study. The purpose of the dose escalation part is to identify the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of CM082 combined with paclitaxel in patients with advanced gastric cancer who did not respond to first-line standard chemotherapy. In the subsequent dose expansion part, additional subjects will be enrolled to further explore the safety and preliminary clinical activity of CM082 and paclitaxel.

DETAILED DESCRIPTION:
In dose escalation part, 9-18 patients with advanced gastric cancer will be enrolled. Patients meeting enrollment eligibility will receive 28-day cycles of CM082 100-200 mg qd combined with paclitaxel 80 mg/m2. Safety information will be collected in cycle 1 to determine MTD and/or RP2D of CM082 combined with paclitaxel in patients with advanced gastric cancer.

Dose escalation study will use traditional 3+3 trial design to observe DLT and evaluate MTD. If there are 2 or more cases of DLT in one dose group, the group lower than this dose group by one level is MTD dose group. At least 6 subjects are required in MTD dose group for confirmation. If MTD is not achieved at the end of dose escalation and there are 6 subjects in the highest dose group, 200 mg qd will be determined as RP2D. Dose escalation and study in the next dose group can be initiated only after the first treatment cycle (DLT window observation period) is completed and safety and tolerability in subject is confirmed in this dose group (0/3 or ≤1/6 subjects experience DLT).

Subjects in the original dose group will continue to receive the next cycle of treatment at the original dose until it meets the following discontinued treatment criteria: 1) death, 2) intolerable toxicity, 3) pregnancy, 4) the investigator considers the study should be terminated for the subject's best interests, 5) the subject or legal representative requests withdrawal, 6) loss to follow-up, 7) the investigator considers the subject has poor compliance, 8) disease progression, 9) the investigator considers the toxicity effect will be intensified if the study continues, 10) use other anti-tumor drugs.

In dose-expansion part, additional patients will be treated at the RP2D established in dose escalation part until it meets the discontinued treatment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and sign the informed consent voluntarily;
* Patients with local advanced and/or metastatic gastric adenocarcinoma and/or adenocarcinoma of gastroesophageal junction confirmed by histology and/or cytology;
* Progressed on previous first-line standard chemotherapy;
* Male or female with an age of 18-70 years(inclusive);
* Body weight ≥40 kg (inclusive);
* At least one measurable lesion (according to RECIST1.1);
* Performance status score (ECOG score) 0-1;
* Expected survival >12 weeks;
* Adequate bonemarrow, liver, renal and cardiac function, based on blood tests, electrocardiograms, and cardiac echocardiograms.

Exclusion Criteria:

* Participating in another drug clinical trial in the past 4 weeks; history of systemic anti-tumor treatment within 4 weeks prior to administration of the study drug; history of any major surgery within 4 weeks prior to enrollment to the study;
* Who have not recovered from toxicity caused by previous anti-cancer treatment (CTCAE>grade 1), or not completely recovered from previous surgery;
* Having received previous chemotherapy regimens with taxanes;
* Take medications that may extend QTc and/or Tdp;
* Active brain metastasis or meningeal metastasis;
* Uncontrolled hypertension (BP>150/90 on medications);
* Other malignancies within the last 5 years, except for adequately treated cervix carcinoma in situ or basal or squamous-cell or basal cell carcinoma;
* QT interval > 450 ms;
* Uncontrolled clinical active infection, e.g. acute pneumonia, active hepatitis B or hepatitis C; HIV positive; syphilitic spiral antibody positive;
* Dysphagia, intractable vomiting or known drug malabsorption;
* Drug or alcohol abuser.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
DLT and MTD | 4 weeks
  DLTs were defined as grade 4 hematological toxicity; grade 3 or more severe nonhematologic toxicity including nausea/vomit, constipation , Hypertension , not controlled by adequate supportive treatment (with exceptions of alopecia); grade 3 febrile neutropenia. The MTD was defined as the highest dose at which no DLT was experienced by the first 3 patients in that cohort, or the dose at which a DLT was experienced by no more than 1 of 6 patients evaluable for toxicity.
Percentage of patients who suffer at least one adverse event | From first dose to within 28 days after the last dose
  Adverse event assessment and changes in safety assessments include laboratory parameters, vital signs, and ECOG score

SECONDARY OUTCOMES:
Objective response rate | 12 weeks
  Defined as the rate of either a complete response or a partial response in evaluable patients
Progression-free survival | 6 months
  Defined as the time from randomisation to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, MD, Study Chair — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided